CLINICAL TRIAL: NCT06634732
Title: Study on the Application Value of Quantitative Ultrasound Assessment Plan for Abdominal Cavity Space in Critically Ill Patients
Brief Title: Quantitative Ultrasound Assessment of Abdominal Cavity Space
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZWQ21886-2024-2
Record Dates: First submitted 2024-09-19; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; MODS; Shock
MeSH Terms: conditions — Sepsis; Multiple Organ Failure; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: Subjectives will undergo abdominal ultrasound examination immediately after receiving an abdominal CT scan.after admission to the ICU.

SUMMARY:
This is a prospective observational study to observe the diagnostic efficacy of a quantitative ultrasound assessment plan for pathological accumulation in the abdominal cavity space of critically ill patients, and to explore its correlation with patient clinical outcomes.

DETAILED DESCRIPTION:
Intra-abdominal lesions, such as hemorrhage and inflammation/infection, often lead to pathological accumulations, posing serious challenges for critically ill patients. These lesions can rapidly induce intra-abdominal hypertension and organ damage, which may progress to hemorrhagic or septic shock, endangering patients' lives. Intra-abdominal hemorrhage, especially surgery-related hemorrhage, is difficult to detect early, and existing assessment methods like CT scans have limited applicability in critically ill patients. Intra-abdominal infections account for a high proportion of infections in critically ill patients, with concurrent sepsis or shock having high mortality rates. Despite advancements in critical care medicine, the mortality rate from intra-abdominal infections remains stubbornly high. Accurate assessment of the source and extent of infection is crucial for treatment, yet routine physical examinations have low sensitivity in critically ill patients, making imaging examinations the primary method. However, while abdominal CT is considered the gold standard, it is limited by insufficient dynamic monitoring and difficulties in patient transport. Bedside ultrasound plays a significant role in the monitoring of critically ill patients due to its portability, non-invasiveness, and real-time dynamic capabilities. It can assess sources of hemorrhage and infection, quantify the extent of lesions, and monitor hemodynamic changes. Therefore, this study aims to develop a comprehensive ultrasound assessment protocol that covers the peritoneal cavity and posterior peritoneal space. Through a prospective observational study, we aim to validate its sensitivity and specificity in diagnosing pathological accumulations such as intra-abdominal hemorrhage/infection and explore its correlation with patient clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;
* Expected ICU stay ≥ 72 hours;
* Meeting one of the diagnostic criteria for intra-abdominal infection: 1) Single organ infection (such as cholecystitis, appendicitis, diverticulitis, cholangitis, pancreatitis, salpingitis, etc.), which may be accompanied by or without peritonitis, even without perforation; 2) Peritonitis, classified as primary, secondary, or recurrent; 3) Intra-abdominal abscess.

Exclusion Criteria:

* Patients with wounds, redness, swelling, bleeding, or other conditions at the abdominal measurement points that prevent ultrasound assessment;
* Patients with intra-abdominal gas accumulation that affects abdominal ultrasound imaging, making ultrasound quantitative scoring impossible;
* Patients who have not undergone abdominal CT examination within 72 hours of ICU admission;
* Patients who do not consent to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in the Department of Critical Care Medicine at Ruijin Hospital, School of Medicine, Shanghai Jiao Tong University
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative CT Scoring for Pathological Accumulations in the Abdominal Cavity Space | up to 3 days after admission to ICU
  score range from 0-20, higher scores indicate a worse outcome
Quantitative Ultrasound Scoring for Pathological Accumulations in the Abdominal Cavity Space | up to 3 days after admission to ICU
  score range from 0-20, higher scores indicate a worse outcome

SECONDARY OUTCOMES:
Time to initiate enteral nutrition | up to 3 days after admission to ICU
  Time to initiate enteral nutrition after admission to ICU in hours
Intra-abdominal pressure | up to 3 days after admission to ICU
  Intra-abdominal pressure in mmHg
C-reactive protein | up to 3 days after admission to ICU
  C-reactive protein in mg/L
procalcitonin | up to 3 days after admission to ICU
  procalcitonin in ng/L
white blood cell count | up to 3 days after admission to ICU
  white blood cell count
time to achieve enteral nutrition targets | up to 28 days after admission to ICU
  time to achieve enteral nutrition targets in hours
serum albumin | up to 28 days after admission to ICU
  serum albumin in g/L
prealbumin | up to 28 days after admission to ICU
  prealbumin in mg/L
Duration of Continuous Renal Replacement Therapy treatment | up to 28 days after admission to ICU
  Duration of CRRT (Continuous Renal Replacement Therapy) treatment in hours
duration of mechanical ventilation | up to 28 days after admission to ICU
  duration of mechanical ventilation in hours
length of ICU stay | up to 28 days after admission to ICU
  length of ICU stay in days
prognosis | up to 28 days after admission to ICU
  survival or death when transfer out of the ICU
acute physiology and chronic health evaluation II score | up to 3 days after admission to ICU
  score range from 0-71, higher scores indicate a worse outcome
Sequential Organ Failure Assessment | up to 3 days after admission to ICU
  score range from 0-15, higher scores indicate a worse outcome
Abdominal Gastrointestinal Index score | up to 3 days after admission to ICU
  score range from 0-4, higher scores indicate a worse outcome
Abdominal Gastrointestinal Index Ultrasonography Score | up to 3 days after admission to ICU
  score range from 0-10, higher scores indicate a worse outcome
Gastrointestinal Ultrasound Scoring score | up to 3 days after admission to ICU
  score range from 0-10, higher scores indicate a worse outcome
semi-quantitative ultrasound score of gastric content | up to 3 days after admission to ICU
  score range from 0-2, higher scores indicate a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided